CLINICAL TRIAL: NCT02693327
Title: Microbiome and the Gut-Brain Axis
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500409
Record Dates: First submitted 2016-02-16; First posted 2016-02-26 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Mental Disorder
Keywords: Gut Microbiome; Mental Disorder; Dysbiosis
MeSH Terms: conditions — Mental Disorders; Dysbiosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mental illness group: Participants in this group will provide biological samples to include both stool and blood samples.
  Interventions: Other: Biological Sample; Other: Blood Sample
- Non-mental illness group: Participants in this group will provide biological samples to include both stool and blood samples.
  Interventions: Other: Biological Sample; Other: Blood Sample

INTERVENTIONS:
Other: Biological Sample — A one time sample will be collected.
  Other Names: Stool Sample
Other: Blood Sample — A one time blood sample will be collected.

SUMMARY:
This research study will examine the relationship interconnecting medical body health, mental health, and microbes of the digestive tract in persons living with serious mental illnesses,as compared to persons without such disorders. Existing research suggests that interactions between digestive tract microbes and the body may influence brain function circuits, mood, anxiety state, cognition, behavior, and medical physiology.

DETAILED DESCRIPTION:
People living with serious mental illnesses have far shorter life expectancy due to various attending medical disorders. Vast knowledge gaps exist regarding microbial taxa responsible for governing various the human states of health or morbidity or interactions with medications. Serious mental illnesses collectively comprise the single largest medical category of life-long disability worldwide. Mounting evidence in humans and in animal models of schizophrenia, post-traumatic stress disorder (PTSD) and related mental illnesses point to gut microbiome-host interactions that may influence brain function circuits, mood, anxiety state, cognition, behavior, as well as generate medical comorbidities. This research study will collect stool samples and blood for in vitro analysis of microbiome and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* People with an existing major mental illness, as already diagnosed currently or within the past year by their doctor prior to being consented,
* Meeting criteria of the fourth or fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV or DSM 5) or ICD-9 or ICD-10;
* Diagnosed with a cardiovascular disorder.

Exclusion Criteria:

* Probiotic use currently or within 2 months prior to study enrollment,
* Antibiotic treatment currently or within 2 months prior to study enrollment;
* Diagnosis of an intellectual disability, pervasive developmental disorder, and/or progressive dementias including Alzheimer's disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1 will have a diagnosis of a mental illness. Group 2 will not have a diagnosis of mental illness.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The potential differences in gut microbiome profiles between persons diagnosed with a major mental illness vs. healthy controls. | Baseline
  In vitro metagenomic sequencing and taxa analyses of gut microbial DNA isolated from stool samples.
Correlation of blood biomarkers with gut microbiome taxa, comparing persons diagnosed with a major mental illness vs. healthy controls. | Baseline
  In vitro analysis of blood biomarkers including short chain fatty acids, inflammatory markers, and evidence for presence of bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R. Stevens, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Department of Medicine, Springhill clinics, Gainesville, Florida
  - Department of Psychiatry, Springhill clinic, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided